CLINICAL TRIAL: NCT02536859
Title: A Randomised, Single-centre, Double-blind, Two-period Cross-over, Multiple Dose Trial Comparing Pharmacodynamic and Pharmacokinetic Properties of Insulin Degludec and Insulin Glargine 300 U/mL at Steady-state Conditions in Subjects With Type 1 Diabetes Mellitus
Brief Title: Comparing Pharmacodynamic and Pharmacokinetic Properties of Insulin Degludec and Insulin Glargine 300 U/mL at Steady-state Conditions in Subjects With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1250-4227; 2014-005602-37 (EudraCT Number); U1111-1165-3940 (Other: WHO)
Record Dates: First submitted 2015-08-28; First posted 2015-09-01 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDeg (Experimental)
  Interventions: Drug: insulin degludec
- IGlar U300 (Active Comparator)
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: insulin degludec — Dose levels will be 0.4 U/kg body weight. The trial products will be administered subcutaneously (s.c., under the skin) once daily.
  Arms: IDeg
Drug: insulin glargine — Dose levels will be 0.4 U/kg body weight. The trial products will be administered subcutaneously (s.c., under the skin) once daily.
  Arms: IGlar U300

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare pharmacodynamic (the effect of the investigated drug on the body) and pharmacokinetic (the exposure of the trial drug in the body) properties of insulin degludec and insulin glargine 300 U/mL at steady-state conditions in subjects with type 1 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-64 years (both inclusive) at the time of signing informed consent
* Subjects diagnosed (clinically) with type 1 diabetes mellitus at least 365 days prior to the day of screening
* Body mass index 18.5-29.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day)who is not able or willing to refrain from smoking or use of nicotine gum or transdermal nicotine patches during the in-patient period

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2016-04-14 (Actual); Study Completion 2016-04-14 (Actual)

PRIMARY OUTCOMES:
Area under the glucose infusion rate curve | During one dosing interval (0-24h) at steady-state. At day 6, 9 and 12

SECONDARY OUTCOMES:
Area under the glucose infusion rate curve | During one dosing interval at steady state.At day 6, 9 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Result] Heise T, Norskov M, Nosek L, Kaplan K, Famulla S, Haahr HL. Insulin degludec: Lower day-to-day and within-day variability in pharmacodynamic response compared with insulin glargine 300 U/mL in type 1 diabetes. Diabetes Obes Metab. 2017 Jul;19(7):1032-1039. doi: 10.1111/dom.12938. Epub 2017 Apr 23. PMID 28295934
- [Result] Heise T, Kaplan K, Haahr HL. Day-to-Day and Within-Day Variability in Glucose-Lowering Effect Between Insulin Degludec and Insulin Glargine (100 U/mL and 300 U/mL): A Comparison Across Studies. J Diabetes Sci Technol. 2018 Mar;12(2):356-363. doi: 10.1177/1932296817731422. Epub 2017 Sep 26. PMID 28946756
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com